CLINICAL TRIAL: NCT06998121
Title: The Effect of Intrarectal Ice Application on Pain, Anxiety, Cortisol Level, Complication Development and Re-admission to Hospital in Transrectal Ultrasonography Guided Prostate Biopsy
Brief Title: The Effect of Intrarectal Ice Application on Pain, Anxiety, Cortisol Level, Complication Development in Transrectal Ultrasonography Guided Prostate Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Elife Kettas Dolek, DR, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MU-001
Record Dates: First submitted 2025-05-29; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Transrectal Ultrasound (TRUS)-Guided Prostate Biopsy
Keywords: Transrectal ultrasound (TRUS)-guided prostate biopsy; intrarectal ice application; pain, anxiety, cortisol levels
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: As a randomised controlled clinical trial, the study population will consist of patients who visit the Urology Outpatient Clinic at Mersin University Hospital and who will undergo transrectal ultrasound-guided prostate biopsy.
Who Masked: Investigator
Masking Description: When it is decided to perform prostate biopsy on patients at the urology outpatient clinic, the researcher (M.B.) will evaluate the patients' eligibility for inclusion in the study. Patients will be assigned to groups using the block randomisation method. Patients will be divided into the study and control groups according to the permutations (ABBA, BABA, etc.) in the randomisation list created by a biostatistician not involved in the study using a computer. After the randomisation list is created, the status of groups A and B as representing the study or control group will be determined by lottery. The coordinating researcher (G.A.U.), who will not be involved in the data collection process of the study, will write numbers from 1 to 96 on the envelope, corresponding to the sample size, and add the letters A or B, representing the groups, inside the envelopes. When the researcher (E.K.D.) visits the patient, they will open the numbered envelope received from the coordinating researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Patients included in the study group will receive intrarectal ice application by researchers (E.K.D. and M.B.) in addition to the outpatient clinic's routine treatment and care practices. For each patient, a new glove (size 8) will be filled with water and frozen to obtain the cold application material. Immediately before the procedure, the lubricated ice will be placed in the patient's rectum and held there for 5 minutes (Caliskan and Mutlu, 2015).
  Pain and anxiety will be assessed in all patients during and after the procedure. At the end of the prostate biopsy, 2 ml of blood will be collected again from the patients to measure serum cortisol levels. The occurrence of complications will be determined by researchers (E.K.D. and G.B.) via telephone during the procedure and one week later. Additionally, when researchers call the patient one week later, they will inquire about any subsequent hospital visits during that period. All information will be recorded on the necessary forms.
  Interventions: Other: Intrarectal ıce application
- contrl (No Intervention): At the outpatient clinic where the study was conducted, oral antibiotic treatment (2x1 Iesef 1 g) was started 24 hours before the prostate biopsy and continued until the dose was completed. A B.T. ENEMA is performed the night before the procedure and at 6:00 a.m. on the day of the procedure. During the procedure, biopsy samples are taken from 12 different areas using a fine needle guided by transrectal ultrasound. Patients who experience pain after the procedure are advised to take oral analgesics (paracetamol). Additionally, patients are informed about precautions to take after the procedure (e.g., seeking medical attention in cases of fever ≥38.5°C and excessive haematuria, avoiding spicy foods for two weeks, etc.). Furthermore, no measures are taken in the outpatient clinic to control pain or anxiety during prostate biopsy. Patients in the control group will receive the outpatient clinic's routine treatment and care.
  Translated with DeepL.com (free version)

INTERVENTIONS:
Other: Intrarectal ıce application — Patients included in the study group will receive intrarectal ice application by researchers (E.K.D. and M.B.) in addition to the outpatient clinic's routine treatment and care practices. For each patient, a new glove (size 8) will be filled with water and frozen to obtain the cold application material. Immediately before the procedure, the lubricated ice will be inserted into the patient's rectum and held in place for 5 minutes (Caliskan and Mutlu, 2015).
  Arms: experimental

SUMMARY:
Transrectal ultrasound (TRUS)-guided prostate biopsy is one of the most commonly performed urological procedures today. This technique involves the insertion of a needle through the rectal mucosa to access the prostate. While TRUS-guided biopsy demonstrates a high detection rate for prostate cancer, it also carries a significant risk of post-procedural complications, such as hematuria, rectal bleeding, urinary retention, and anemia.

Compared to other biopsy methods, TRUS-guided biopsy is associated with higher rates of hospital readmissions and an increased risk of infection and sepsis. These complications contribute to elevated healthcare costs, prolonged hospital stays, increased workload for healthcare providers, heightened patient stress and anxiety levels, greater analgesic requirements, the potential for additional complications, and reduced patient satisfaction.

Various non-pharmacological methods have been shown to be effective in preventing these adverse patient outcomes. One such method, which has been identified in the literature as effective, is cold application. Cold application is a widely preferred non-pharmacological intervention due to its simplicity, affordability, and accessibility. It is particularly used to reduce acute pain, edema, and bleeding. Cold therapy slows down metabolism, thereby reducing the oxygen and nutrient demands of tissues; it also limits inflammation, muscle spasm, and edema, alleviates pressure and tension on nerve endings, and decreases the conduction velocity of peripheral nerves. These effects contribute to a reduction in patients' pain, anxiety associated with pain, and bleeding.

The aim of this study is to determine the effects of intrarectal ice application during transrectal ultrasound-guided prostate biopsy on pain, anxiety, cortisol levels, the incidence of complications, and hospital readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study,
* Patients over the age of 18
* Patients who are conscious, oriented, and cooperative,
* Patients who have no communication problems,
* Patients who are scheduled to undergo their first prostate biopsy under transrectal ultrasound guidance,
* Patients who have no mental disorders,
* Patients who have not been diagnosed with anxiety disorder,
* Patients not taking medication for anxiety control.

Exclusion Criteria:

* Patients who refuse to participate in the study,
* Patients under the age of 18
* Patients who are conscious, oriented, and uncooperative,
* Patients with communication problems,
* Patients who have not undergone transrectal ultrasound-guided prostate biopsy,
* Patients who have previously undergone prostate biopsy,
* Patients with mental disorders,
* Patients diagnosed with anxiety disorder,
* Patients taking medication for anxiety control.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The procedure is specific to men because a prostate biopsy will be performed.
Enrollment: 84 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 12 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Pain score | 12 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).
Patient Outcomes | 12 months
  Patient Follow-up Form: This form will record patients' serum cortisol levels before and after the biopsy procedure, complications that develop within one week after the biopsy (rectal bleeding, haematuria, urinary retention, anaemia, infection, etc.) and whether the patient returns to the hospital during this period.